CLINICAL TRIAL: NCT02703428
Title: The LUCY Study: TriVascular Evaluation of Females Who Are Underrepresented Candidates for Abdominal Aortic Aneurysm Repair in Europe
Brief Title: TriVascular Evaluation of Females Who Are Underrepresented Candidates for Abdominal Aortic Aneurysm Repair in Europe
Acronym: LUCY
Status: Completed | Type: Observational
Sponsor: TriVascular, Inc. (Industry)
Collaborators: Endologix (Industry)
Responsible Party: Sponsor
Organization: Endologix (Industry)
Other Study IDs: 771-0019
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal; Aortic; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The LUCY Study is a prospective, consecutively enrolling, non-randomized multi center post-market study to evaluate the low profile (14F) Ovation® Abdominal Stent Graft Platform when used in the endovascular treatment of female patients.

DETAILED DESCRIPTION:
The LUCY Study is a prospective, consecutively enrolling, non-randomized multi center post-market study to evaluate the Ovation Abdominal Platform when used in the endovascular treatment of female patients.

The primary endpoint is freedom from access-related vascular complications and freedom from AAA-related mortality through 30 days.

Secondary endpoints of the study will be achieved by demonstrating the benefits in female patients despite the fact that historically fewer female patients have been eligible for EVAR, and they have experienced a higher rate of access-related complications and higher mortality rates. Secondary endpoints will be evaluated through 1 year (365 ± 60 days) post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age.
2. Patients who are non-pregnant female (females of child bearing potential must have a negative pregnancy test prior to enrollment into the study).
3. Patient has signed an Ethics Committee (EC) approved Informed Consent Form.
4. Patient is considered by the treating physician to be a candidate for elective open surgical repair of the AAA (i.e., category I, II, or III per American Society of Anesthesiology (ASA) classification). ASA category IV patients may be enrolled provided their life expectancy is greater than 1 year.
5. Patient has an infrarenal abdominal aortic aneurysm that meets at least one of the following:

   * Abdominal aortic aneurysm >5.0 cm in diameter;
   * Aneurysm has increased in size by 0.5 cm in last 6 months; or
   * Maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent non-aneurysmal aortic segment.
6. Patient has suitable anatomy that allows use of the TriVascular Ovation Abdominal Platform:

   * Iliac or femoral arteries that allow endovascular access with the TriVascular Ovation Abdominal Platform.
   * Proximal aortic neck landing zone with an inner wall diameter of no less than 16 mm and no greater than 30 mm at 13 mm below the inferior renal artery.
   * Distal iliac artery landing zone length (seal zone) of ≥10 mm. The resultant repair should preserve patency in at least one hypogastric artery.
   * Distal iliac artery landing zone an inner wall diameter of no less than 8 mm and no greater than 25 mm.
   * Distance from the most distal renal artery to most superior internal iliac artery measurement is at least 130 mm.
   * Aortic angle of ≤ 60 degrees if proximal neck length is ≥10 mm and ≤ 45 degrees if proximal neck length is <10 mm.
7. Patient must be willing to comply with all required follow-up exams.

Exclusion Criteria:

1. Patient has a need for emergent surgery.
2. Patient has a dissecting aneurysm.
3. Patient has an acutely ruptured aneurysm.
4. Patient has an acute vascular injury.
5. Patient has had a previous repair of the abdominal aortic aneurysm or an iliac artery in intended treatment zone.
6. Patient has a known thoracic aortic aneurysm or dissection that will require treatment (surgery or endovascular intervention) within the study period.
7. Patient has a mycotic aneurysm or has an active systemic infection.
8. Patient has unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina, or onset of prolonged angina).
9. Patient has had a myocardial infarction (MI) and/or stroke (CVA) within the past 6 months.
10. Patient requires use of techniques (e.g. Chimney graft) that would cover the renal arteries.
11. Patient requires planned adjunctive devices (e.g. renal stents) to complete the procedure.
12. Patient has a major surgical or interventional procedure planned during or within ±30 days of the AAA repair.
13. Patient has history of connective tissue disease (e.g., Marfan's or Ehler's-Danlos syndrome).
14. Patient has history of bleeding disorders or refuses blood transfusions.
15. Patient has dialysis dependent renal failure or baseline serum creatinine level >2.0 mg/dl
16. Patient has a known hypersensitivity or contraindication to anticoagulation or contrast media that is not amenable to pre-treatment.
17. Patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE), PEG-based polymers, fluorinated ethylene propylene (FEP) or nitinol.
18. Patient has a body habitus that would inhibit X-ray visualization of the aorta.
19. Patient has a limited life expectancy of less than 1 year.
20. Patient is currently participating in an investigational device or drug clinical trial.
21. Patient has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll female subjects, 18 years of age or older that have an AAA and meet all other inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Freedom from access-related vascular complications and freedom from AAA-related mortality through 30 days. | 30 ± 10 days

SECONDARY OUTCOMES:
Serious and Non-Serious Adverse Events | 365 ± 60 days
Access-related vascular complications | 365 ± 60 days
Technical (deployment) success | 365 ± 60 days
  Defined as successful delivery and deployment of one aortic body and at least two iliac limbs.
Freedom from Type I & III endoleaks | 365 ± 60 days
Freedom from migration | 365 ± 60 days
Freedom from aneurysm enlargement | 365 ± 60 days
Freedom from Abdominal Aortic Aneurysm rupture | 365 ± 60 days
Freedom from conversion to open repair | 365 ± 60 days
  Conversion to open surgical repair occurs when a subject implanted with an Ovation Abdominal Platform undergoes open surgical repair with explantation of the stent graft.
Freedom from AAA related secondary interventions | 365 ± 60 days
Freedom from mortality (all cause and AAA related) | 365 ± 60 days
Blood Loss | 365 ± 60 days
  Estimate blood loss and replacement requirements, (e.g. transfusion).
Duration of Procedure | 365 ± 60 days
  Time enter procedure room, time start arterial access, stent graft deployment start and stop time, time of closure of arterial access, and time exit procedure room.
Length of hospital and ICU (if required) | 365 ± 60 days
Anesthesia Type | 365 ± 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kolvenbach, M.D., Ph.D., Principal Investigator — Augusta Krankenhaus
Locations (10):
- Belgium (2):
  - OLV Ziekhenuis, Aalst
  - UZ Leuven, Leuven
- Germany (6):
  - HGZ Bad Bevensen, Bad Bevensen
  - August Krankenhaus, Düsseldorf
  - University of Düsseldorf, Düsseldorf
  - University Medical Center Hamburg, Hamburg
  - Hospital Karlsruhe, Karlsruhe
  - University of Leipzig, Leipzig
- Institute of Hematology and Blood Transfusion, Warsaw, Poland
- Bedfordshire Hospitals NHS Trust, Bedford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.endologix.com